CLINICAL TRIAL: NCT05663723
Title: Photobiomodulation for Prevention of Chemotherapy-induced Peripheral Neuropathy in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erica Alves Nogueira Fabro (Other Government)
Collaborators: COSMEDICAL (Unknown); BLED MED COMERCIO E DISTRIBUIÇÃO LTDA (Unknown)
Responsible Party: Sponsor-Investigator, Erica Alves Nogueira Fabro, Technical manager, Instituto Nacional de Cancer, Brazil
Organization: Instituto Nacional de Cancer, Brazil (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Prevention of neuropathy
Record Dates: First submitted 2022-11-30; First posted 2022-12-23 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Nervous System Diseases AND Breast Neoplasms
Keywords: Breast cancer; Peripheral neuropathy; Chemotherapy; Photobiomodulation
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The intervention and control groups will be: Group A: Intervention group with the IV and V LED board. Group B: Intervention group with the IV, V and Violet LED board. Group C: Control group with the LED board without emitting light.
Who Masked: Participant, Outcomes Assessor
Masking Description: Only outcome assessors and patients will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group with the IV and V LED board (Active Comparator): Time of Applications will for 20 minutes on each extremity (foot soles), until the last day of chemotherapy treatment. The sequential LED treatments will be administered by the Sportllux Ultra model (Cosmedical) in a predefined cycle, with the combination of light emitters in two wavelengths: 42 red (660nm) and 42 infrared (850nm); LED blanket in the size of 10x12 cm; average power of each LED: 5mW; operating mode: continuous; polarization: random; irradiance at the opening of each LED: 25mW/cm2; opening diameter of each LED: 10mm; application time: 1 session of 20 minutes; power per LED: 30mW; radiant exposure: 36J/cm2 during 20 minutes of application. Tissue from the lower limb extremities will come into contact with the LED panel during treatment to ensure even delivery of photobiomodulation. The panels are large enough to more than cover the entire edge area at one time during application.
  Interventions: Device: Intervention group with the IV and V LED board
- Intervention group with the IV, V and Violet LED board (Active Comparator): Time of Applications will be for 20 minutes on each extremity (foot soles), until the last day of chemotherapy treatment. The sequential LED treatments will be administered by the Sportllux Ultra model (Cosmedical) in a predefined cycle, with the combination of light emitters in three wavelengths: 18 red (660nm), 18 infrared (850nm) and 36 violet (420nm). ); LED blanket in the size of 10x12 cm; average power of each LED: 5mW; operating mode: continuous; polarization: random; irradiance at the opening of each LED: 25mW/cm2; opening diameter of each LED: 10mm; application time: 1 session of 20 minutes; power per LED: 30mW; radiant exposure: 36J/cm2 during 20 minutes of application. Tissue from the lower limb extremities will come into contact with the LED panel during treatment to ensure even delivery of photobiomodulation. The panels are large enough to more than cover the entire edge area at one time during application.
  Interventions: Device: Intervention group with the IV, V and Violet LED board
- Control group with LED board without emitting light (Placebo Comparator): Applications of the LED board will be performed daily for 20 minutes on each extremity (foot soles), until the last day of chemotherapy treatment. The sequential LED treatments will be administered by the Sportllux Ultra (Cosmedical) model without the light emitting combination. LED blanket in the size of 10x12 cm and application time: 1 session of 20 minutes. Tissue from the lower limb extremities will come into contact with the LED panel during treatment to ensure even delivery of photobiomodulation. The panels are large enough to more than cover the entire edge area at one time during application. Women will receive a booklet with guidelines for the correct use of the LED board and will be instructed to continue their usual physical activities and mark the daily frequency of application of the LED board
  Interventions: Device: Control group with LED board without emitting light

INTERVENTIONS:
Device: Intervention group with the IV and V LED board — Applications of the LED board will be performed daily for 20 minutes on each extremity (foot soles), until the last day of chemotherapy treatment. The sequential LED treatments will be administered by the Sportllux Ultra model (Cosmedical) in a predefined cycle, with the combination of light emitters in two wavelengths: 42 red (660nm) and 42 infrared (850nm); LED blanket in the size of 10x12 cm; average power of each LED: 5mW; operating mode: continuous; polarization: random; irradiance at the opening of each LED: 25mW/cm2; opening diameter of each LED: 10mm; application time: 1 session of 20 minutes; power per LED: 30mW; radiant exposure: 36J/cm2 during 20 minutes of application. Tissue from the lower limb extremities will come into contact with the LED panel during treatment to ensure even delivery of photobiomodulation. The panels are large enough to more than cover the entire edge area at one time during application.
  Arms: Intervention group with the IV and V LED board
Device: Intervention group with the IV, V and Violet LED board — Applications of the LED board will be performed daily for 20 minutes on each extremity (foot soles), until the last day of chemotherapy treatment. The sequential LED treatments will be administered by the Sportllux Ultra model (Cosmedical) in a predefined cycle, with the combination of light emitters in three wavelengths: 18 red (660nm), 18 infrared (850nm) and 36 violet (420nm). ); LED blanket in the size of 10x12 cm; average power of each LED: 5mW; operating mode: continuous; polarization: random; irradiance at the opening of each LED: 25mW/cm2; opening diameter of each LED: 10mm; application time: 1 session of 20 minutes; power per LED: 30mW; radiant exposure: 36J/cm2 during 20 minutes of application. Tissue from the lower limb extremities will come into contact with the LED panel during treatment to ensure even delivery of photobiomodulation. The panels are large enough to more than cover the entire edge area at one time during application.
  Arms: Intervention group with the IV, V and Violet LED board
Device: Control group with LED board without emitting light — Applications of the LED board will be performed daily for 20 minutes on each extremity (foot soles), until the last day of chemotherapy treatment. The sequential LED treatments will be administered by the Sportllux Ultra (Cosmedical) model without the light emitting combination. LED blanket in the size of 10x12 cm and application time: 1 session of 20 minutes. Tissue from the lower limb extremities will come into contact with the LED panel during treatment to ensure even delivery of photobiomodulation. The panels are large enough to more than cover the entire edge area at one time during application.
  Arms: Control group with LED board without emitting light

SUMMARY:
Double-blind Superiority Randomized Controlled Clinical Trial. Objective of the study: To evaluate the effectiveness of photobiomodulation using the LED board in the prevention of peripheral neuropathy in the lower limbs in women with breast cancer undergoing chemotherapy at the Cancer Hospital III of the National Cancer Institute (HCIII/INCA).

DETAILED DESCRIPTION:
Materials and methods: This is a single-blind superiority randomized controlled clinical trial. Women aged over 18 years, with breast cancer in stages I to IIIC and who have an indication for curative treatment with neoadjuvant or adjuvant chemotherapy at HCIII/INCA will be eligible. Patients with a previous diagnosis of another primary cancer will be excluded; patients undergoing surgery and/or chemotherapy at another institution; patients who previously had altered sensitivity in the feet; patients who are unable to answer the questionnaires and patients unable to receive photobiomodulation due to acute infections in the lower limbs. After recruitment, the women will be allocated into three groups: two Intervention groups (use of the IV and V LED board; and IV, V and Violet) and a Control group (use of the LED board without light emission). Peripheral neuropathy, pain, global muscle strength, body balance, sensitivity, health-related quality of life and related independent variables will be evaluated, such as the characteristics of the patient, the tumor and the oncological treatment performed. Data analysis: Statistical analysis will be conducted following intention-to-treat principles. Data normality will be tested using the Kolmogorov Smirnov test, considering as normal distribution those with p > 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Women aged over 18 years, with breast cancer in stages I to IIIC and who have an indication for curative treatment with neoadjuvant or adjuvant chemotherapy in HCIII/INCA.

Exclusion Criteria:

* Patients with a previous diagnosis of another primary cancer
* Patients undergoing surgery and/or chemotherapy at another Institution
* Patients who previously had altered sensitivity in the feet
* Patients who are unable to respond to questionnaires
* Patients unable to receive photobiomodulation due to acute lower limb infections

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women diagnosed with breast cancer
Enrollment: 186 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Peripheral neuropathy | Until the conclusion of the study, on average 14 months
  Chemotherapy Induced Peripheral Neuropathy Assessment Tool (FANPIQ), which is validated and translated from the Chemotherapy Induced Peripheral Neuropathy Assessment Tool - (CIPNAT).

SECONDARY OUTCOMES:
Lower limb pain | Until the conclusion of the study, on average 14 months
  Short Form McGill Questionnaire, which is the McGill questionnaire in its shortened form
Overall Muscle Strength | Until the conclusion of the study, on average 14 months
  Hydraulic Jamar Dynamometer (Sammons Preston Rolyan, 4, Sammons Court, Bolingbrook, IL, 60440)
Body Balance | Until the conclusion of the study, on average 14 months
  Timed Up and Go Test (TUG)
Lower limb sensitivity | until the conclusion of the study, on average 14 months
  Esthesiometer (monofilaments)
Health-related quality of life | Until the conclusion of the study, on average 14 months
  Functional Assessment of Cancer Therapy/Gynaecologic Oncology Group - Neurotoxicity Questionnaire (FACT/GOG-NTX), Portuguese version FACT/GOG-NTX (Portuguese version)
Satisfaction with the use of photobiomodulation | Until the conclusion of the study, on average 14 months
  Questions will be asked about overall satisfaction with the management of peripheral neuropathy
Assessment of Adherence to Treatment | Until the conclusion of the study, on average 14 months
  The LED board application diary will be used in which patients in intervention group A and B and control will be instructed to fill it in daily during the intervention period. In this diary, patients must inform the date of application of the LED board, if it was performed on both feet and if the duration time was 20 minutes on each limb. The LED board application diary must be delivered by the patient or family member to a physiotherapist who will be responsible for receiving it, on the last day of the chemotherapy treatment.
Impact of Peripheral Neuropathy on Activities of Daily Living | Until the conclusion of the study, on average 14 months
  Chemotherapy Induced Peripheral Neuropathy Assessment Tool (FANPIQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Erica Alves Nogueira Fabro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrade, L.C.A; Costa G.L.A. and other Timed Up and Go test in assessing the risk of falls in the elderly: a literature review. Research, Society and Development. 2021, 10(13):1-7.
- [Background] Alberto, Talita; Corbo, B.F.B; e outros Efeitos do emissor de luz (LED) vermelho na estimulação de fibroblastos: ansiedade na emoção tecidual. Revista Intellectus. Vol 1, n. 33 de 2016.
- [Background] Andreo L, Soldera CB, Ribeiro BG, de Matos PRV, Bussadori SK, Fernandes KPS, Mesquita-Ferrari RA. Effects of photobiomodulation on experimental models of peripheral nerve injury. Lasers Med Sci. 2017 Dec;32(9):2155-2165. doi: 10.1007/s10103-017-2359-7. Epub 2017 Oct 23. PMID 29063472
- [Background] Argenta PA, Ballman KV, Geller MA, Carson LF, Ghebre R, Mullany SA, Teoh DG, Winterhoff BJ, Rivard CL, Erickson BK. The effect of photobiomodulation on chemotherapy-induced peripheral neuropathy: A randomized, sham-controlled clinical trial. Gynecol Oncol. 2017 Jan;144(1):159-166. doi: 10.1016/j.ygyno.2016.11.013. Epub 2016 Nov 22. PMID 27887804
- [Background] Rafael Inácio Barbosa, R.I; Marcolino A.M; Guirro R.R.J; Nilton Mazzer, Nilton; et al. Efeito do laser de baixa intensidade (660 nm) na regeneração do nervo isquiático lesado em ratos. Fisioterapia e Pesquisa, São Paulo, v.17, n.4, p. 294-9, out/dez. 2010.
- [Background] Bensadoun RJ, Bollet MA, Liem X, Cao K, Magne N. New photobiomodulation device for prevention and cure of radiotherapy-induced oral mucositis and dermatitis: results of the prospective Safe PBM study. Support Care Cancer. 2022 Feb;30(2):1569-1577. doi: 10.1007/s00520-021-06574-2. Epub 2021 Sep 19. PMID 34537889
- [Background] Bethesda, MD: National Cancer Institute. PDQ® Adult Treatment Editorial Board. PDQ Breast Cancer Treatment (Adult). Available at: https://www.cancer.gov/types/breast/hp/breast-treatment-pdq. Accessed August 10th, 2022.
- [Background] Brasil. Ministério da Saúde; Instituto Nacional de Câncer José Alencar Gomes da Silva. Ações de enfermagem para o controle do câncer: uma proposta de integração ensino-serviço. Rio de Janeiro: INCA; 2008. Bases do tratamento; p. 369-556.
- [Background] Beliche T.W.O; Hamu T.C.D.S. et al. Diferenças de aplicação do teste timed up and go em crianças típicas. Revista Temas em Saúde, v. 20, n°1, p. 95-103. João Pessoa,2020.
- [Background] Bretan O, Silva Junior JE, Ribeiro OR, Corrente JE. Risk of falling among elderly persons living in the community: assessment by the Timed up and go test. Braz J Otorhinolaryngol. 2013 Jan-Feb;79(1):18-21. doi: 10.5935/1808-8694.20130004. PMID 23503902
- [Background] Calhoun EA, Welshman EE, Chang CH, Lurain JR, Fishman DA, Hunt TL, Cella D. Psychometric evaluation of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (Fact/GOG-Ntx) questionnaire for patients receiving systemic chemotherapy. Int J Gynecol Cancer. 2003 Nov-Dec;13(6):741-8. doi: 10.1111/j.1525-1438.2003.13603.x. PMID 14675309
- [Background] Costa TC, Lopes M, Anjos AC, Zago MM. [Chemotherapy-induced peripheral neuropathies: an integrative review of the literature]. Rev Esc Enferm USP. 2015 Apr;49(2):335-45. doi: 10.1590/S0080-623420150000200020. Portuguese. PMID 25992834
- [Background] DUTRA M. C; CABRAL A. L. L, CARVALHO G. A. Tradução para o português e validação do teste timed up and go. Revista Interfaces. Saúde, Humanas e Tecnologia. Vol. 3(9), pp. 81-88, 22 de Abril, 2016
- [Background] Fisusi FA, Akala EO. Drug Combinations in Breast Cancer Therapy. Pharm Nanotechnol. 2019;7(1):3-23. doi: 10.2174/2211738507666190122111224. PMID 30666921
- [Background] Fernandes A.A; Marins J.C.B. Teste de força de preensão manual: análise metodológica e dados normativos em atletas. Fisioter. mov. 24 (3). Set 2011.
- [Background] Heiskanen V, Hamblin MR. Photobiomodulation: lasers vs. light emitting diodes? Photochem Photobiol Sci. 2018 Aug 8;17(8):1003-1017. doi: 10.1039/c8pp90049c. PMID 30044464
- [Background] Hsieh YL, Fan YC, Yang CC. Low-level laser therapy alleviates mechanical and cold allodynia induced by oxaliplatin administration in rats. Support Care Cancer. 2016 Jan;24(1):233-242. doi: 10.1007/s00520-015-2773-y. Epub 2015 May 26. PMID 26006084
- [Background] Instituto Nacional de Câncer José Alencar Gomes da Silva. Estimativa 2020: incidência de câncer de mama no Brasil. Rio de Janeiro: INCA; 2021. [acesso em agosto 2021]. Disponível: http://www.inca.gov.br.
- [Background] LEHMAN, L. F. et al. Avaliação neurológica simplificada. Belo Horizonte: ALM International, 1997. 104 p.
- [Background] Joy L, Jolien R, Marithe C, Stijn E, Laura S, Hilde L, Sandra B, Wendy N, Ruth H, Liesbeth R, Sylvana S, Sylvia H, Jeroen M. The use of photobiomodulation therapy for the prevention of chemotherapy-induced peripheral neuropathy: a randomized, placebo-controlled pilot trial (NEUROLASER trial). Support Care Cancer. 2022 Jun;30(6):5509-5517. doi: 10.1007/s00520-022-06975-x. Epub 2022 Mar 21. PMID 35312857
- [Background] Lodewijckx J, Robijns J, Bensadoun RJ, Mebis J. Photobiomodulation Therapy for the Management of Chemotherapy-Induced Peripheral Neuropathy: An Overview. Photobiomodul Photomed Laser Surg. 2020 Jun;38(6):348-354. doi: 10.1089/photob.2019.4771. Epub 2020 May 28. PMID 32460667
- [Background] Malta CEN, Carlos ACAM, de Alencar MCM, Alves E Silva EF, Nogueira VBC, Alves APNN, Chaves FF, de Moura JFB, de Barros Silva PG. Photobiomodulation therapy prevents dysgeusia chemotherapy induced in breast cancer women treated with doxorubicin plus cyclophosphamide: a triple-blinded, randomized, placebo-controlled clinical trial. Support Care Cancer. 2022 Mar;30(3):2569-2580. doi: 10.1007/s00520-021-06642-7. Epub 2021 Nov 19. PMID 34799776
- [Background] Martin LG, Silva MD. Chemotherapy-induced peripheral neuropathy: a literature review. Einstein (Sao Paulo). 2011 Dec;9(4):538-44. doi: 10.1590/S1679-45082011RW2220. English, Portuguese. PMID 26761262
- [Background] Martinez B.P; Santos M. R; et al. SEGURANÇA E REPRODUTIBILIDADE DO TESTE TIMED UP AND GO EM IDOSOS HOSPITALIZADOS. Rev Bras Med Esporte - Vol. 22, No 5 - Set/Out, 2016.
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Pereira, Esdras Edgar Batista; SANTOS, Nadia Barreto dos; SARGES, Edilene do Socorro Nascimento Falcão. Avaliação da capacidade funcional do paciente oncogeriátrico hospitalizado. Revista Pan-Amazônica de Saúde, v. 5, n. 4, p. 37-44, 2014.
- [Background] Reis, Mariana Xavier. Escalas de Avaliação de Neuropatia Periférica Induzida por Quimioterapia - Uma revisão. São Luiz,2016.
- [Background] Rezende,L; Campanholi, LL; Tessaro, A. Manual de Condutas e Práticas Fisioterapêuticas no Câncer de Mama da ABFO. 1 ed. Rio de Janeiro; Thieme Revinter Publicações, 2018.
- [Background] Sene GA, Sousa FF, Fazan VS, Barbieri CH. Effects of laser therapy in peripheral nerve regeneration. Acta Ortop Bras. 2013;21(5):266-70. doi: 10.1590/S1413-78522013000500005. PMID 24453680
- [Background] Shien T, Iwata H. Adjuvant and neoadjuvant therapy for breast cancer. Jpn J Clin Oncol. 2020 Mar 9;50(3):225-229. doi: 10.1093/jjco/hyz213. PMID 32147701
- [Background] Simão, DAS. Estudo da neuropatia periférica induzida por quimioterapia: possíveis preditores clínicos e validação de instrumento de avaliação, 2015.
- [Background] Simão, D.A.S.; Murad, M.; et al. Neuropatia periférica induzida por quimioterapia: revisão para a prática clínica. Rev Dor. São Paulo, 2015 jul-set;16(3):215-20.
- [Background] Simão, D.A.S; Abreu, M.N.S; Gomez, R.S; et al. Evolução Clínica e Preditores da Neuropatia Periférica Induzida por Quimioterapia. Revista Brasileira de Cancerologia 2019; 65(2): e-04392.
- [Background] da Silva Simao DA, Teixeira AL, Souza RS, de Paula Lima ED. Evaluation of the Semmes-Weinstein filaments and a questionnaire to assess chemotherapy-induced peripheral neuropathy. Support Care Cancer. 2014 Oct;22(10):2767-73. doi: 10.1007/s00520-014-2275-3. Epub 2014 May 9. PMID 24811218
- [Background] Souza, FN. Avaliação da dor em pacientes oncológicos em um hospital escola da cidade de Florianópolis/SC. Florianópolis, SC, 2020.
- [Background] Zandonai, AP. Adaptação transcultural e validação do instrument Chemotherapy-Induced Peripheral Neuropathy Assessment Tool (CIPNAT) para o Brasil. Tese de Doutorado, apresentada à Escola de Enfermagem de Ribeirão Preto/USP. Área de concentração: Enfermagem Fundamental. Ribeirão Preto,2015.
- [Background] Zecha JA, Raber-Durlacher JE, Nair RG, Epstein JB, Elad S, Hamblin MR, Barasch A, Migliorati CA, Milstein DM, Genot MT, Lansaat L, van der Brink R, Arnabat-Dominguez J, van der Molen L, Jacobi I, van Diessen J, de Lange J, Smeele LE, Schubert MM, Bensadoun RJ. Low-level laser therapy/photobiomodulation in the management of side effects of chemoradiation therapy in head and neck cancer: part 2: proposed applications and treatment protocols. Support Care Cancer. 2016 Jun;24(6):2793-805. doi: 10.1007/s00520-016-3153-y. Epub 2016 Mar 17. PMID 26984249
- [Background] Wamser E.L, Valderramas S.R, Paula J.Á. Et al. Melhor Desempenho no teste Timed Up And Go está associado a melhor desempenho funcional em idosas da comunidade. Geriatr Gerontol Aging. 2015; 9(4):138-43.
- [Background] Wang Y, Ge Y, Xing W, Liu J, Wu J, Lin H, Lu Y. The effectiveness and safety of low-level laser therapy on breast cancer-related lymphedema: An overview and update of systematic reviews. Lasers Med Sci. 2022 Apr;37(3):1389-1413. doi: 10.1007/s10103-021-03446-3. Epub 2021 Nov 15. PMID 34779937